CLINICAL TRIAL: NCT01094899
Title: Study of Abnormal Structure and Bone Density at the Feet of Diabetic Patients
Brief Title: Abnormal Structure and Bone Density in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C08-25; 2008-A00937-48 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-03-10; First posted 2010-03-29 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: diabetes; osteopenia; neuropathy; foot; AGE
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Bone Diseases, Metabolic | interventions — X-Rays; Urination; Blood Specimen Collection; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Type 1 Diabetics without Neuropathy (Experimental): Adult male with type 1 diabetes and without peripherical neuropathy
  Interventions: Radiation: Radiography; Other: Urine and Blood sampling; Other: Echography
- Type 2 Diabetics without Neuropathy (Experimental): Adult male with type 2 diabetes and without peripherical neuropathy
  Interventions: Radiation: Radiography; Other: Urine and Blood sampling; Other: Echography
- Type 1 Diabetics with Neuropathy (Experimental): Adult male with type 1 diabetes and with peripherical neuropathy
  Interventions: Radiation: Radiography; Other: Urine and Blood sampling; Other: Echography
- Type 2 Diabetics with Neuropathy (Experimental): Adult male with type 1 diabetes and with peripherical neuropathy
  Interventions: Radiation: Radiography; Other: Urine and Blood sampling; Other: Echography

INTERVENTIONS:
Radiation: Radiography — Radiography, microscanner, osteodensitometry
Other: Urine and Blood sampling — mainly dosage of bones metabolism
Other: Echography — body bones echography

SUMMARY:
Assumptions and Objectives: The working hypotheses are: 1 - subjects with type 1 diabetes and / or type 2, compared to subjects without diabetes are at risk for osteopenia and / or abnormal bone structure the foot (calcaneus and ankle) can lead to bone deformities, fractures and final stage of Charcot foot. These anomalies are favored by the presence of peripheral neuropathy and plasma levels of advanced glycation end products higher than in diabetic subjects without bone abnormalities.

The objectives of this research are to evaluate these anomalies quantitative and qualitative bone in the foot (calcaneus and ankle) through the use of MicroScanner. In parallel a whole body bone mineral density (BMD) and calcaneal ultrasound will be performed to measure bone mineral density as realized in clinical practice in a defined population of patients with type 1 or type 2. These bone abnormalities will be correlated with the presence of peripheral neuropathy and the rate of advanced glycation end products of proteins and reference to parameters of chronic inflammation and oxidative stress to better understand the pathophysiology and target a population at risk.

The importance of this study is paramount in the management of diabetic foot. Indeed for the moment we are dealing primarily the consequences of diabetes impact bone when bone deformities have appeared with their attendant disability and the risk of recurrent infections in areas of friction in this fragile environment. The ultimate goal is to target people with diabetes have abnormal bone subclinical and take care to avoid changes to bone deformities and find ways to treat them.

DETAILED DESCRIPTION:
The population studies on subjects with type 1 and 2 diabetes have revealed a fracture risk multiplied by 4 to 12, especially at the shoulder, hip, ankle and foot, compared to a population of non-diabetic subjects matched for age and sex.

If osteopenia (decreased bone mineral density) is consistently associated with fracture risk in diabetic patients with type 1 diabetes type 2 often have a bone mineral density comparable or superior to non diabetes subjects.

The various causes mentioned in this alteration of the quantity and bone quality in the context of chronic hyperglycemia is a disturbance of the interaction between osteoblasts (cells forming bone) and osteoclasts (cells that resorb bone), partly mediated by the system RANK / RANK-L / osteoprotegerin with decreased bone formation and increased osteolyses. The peripherical neuropathy, the glycation proteins (modifications of proteins by addition of glucose) and the receptor of glycation proteins are directly involved.

At the foot, these changes in the bones (osteopenia and decreased bone quality) are responsible for deformations observed in some diabetic subjects, resulting in the formation of "Charcot foot" and the risk of sores and amputation as a major disability cause. Few studies have examined the abnormalities that we could find at the foot of the diabetic patients before the development of deformities observed in the Charcot foot. One study looked at bone mineral density measured by ultrasound at the Charcot foot and the contralateral foot in subjects with type 1 or type 2 compared to subjects with no diabetic Charcot foot. The authors found a decrease in bone density measured by ultrasound at the Charcot foot compared with the contralateral foot in subjects with type 1 and type 2. Bone density at the contralateral foot was reduced compared with control subjects with diabetes only in subjects with type 1 diabetes but not in patients with type 2 diabetes. The link with the peripheral neuropathy is not clear. A second study in women with type 1 diabetes in premenopausal also found a decrease in bone density at the calcaneus measured by ultrasound compared with women without diabetes. None of these studies focused on the local structure of the bone. Yet we may suspect that hyperglycemia, including glycation of proteins may cause structural changes in the bone of diabetic subjects. Previously, it was difficult to understand the structure of bone by non-invasive, the MicroScanner developed by the Scanco company can measure bone density and trabecular architecture of the wrist and ankle with a discrimination of 42 microns . He does a minimal radiation (3 microsV) and allows a resolution of 80 microns. It has already been used in osteopenic women and showed significant differences in terms of bone architecture between women with fracture and those who do not.

Assumptions and Objectives: The working hypotheses are: 1 - subjects with type 1 diabetes and / or type 2, compared to subjects without diabetes are at risk for osteopenia and / or abnormal bone structure the foot (calcaneus and ankle) can lead to bone deformities, fractures and final stage of Charcot foot. These anomalies are favored by the presence of peripheral neuropathy and plasma levels of advanced glycation end products higher than in diabetic subjects without bone abnormalities.

The objectives of this research are to evaluate these anomalies quantitative and qualitative bone in the foot (calcaneus and ankle) through the use of MicroScanner. In parallel a whole body BMD and calcaneal ultrasound will be performed to measure bone mineral density as realized in clinical practice in a defined population of patients with type 1 or type 2. These bone abnormalities will be correlated with the presence of peripheral neuropathy and the rate of advanced glycation end products of proteins and reference to parameters of chronic inflammation and oxidative stress to better understand the pathophysiology and target a population at risk.

The importance of this study is paramount in the management of diabetic foot. Indeed for the moment we are dealing primarily the consequences of diabetes impact bone when bone deformities have appeared with their attendant disability and the risk of recurrent infections in areas of friction in this fragile environment. The ultimate goal is to target people with diabetes have abnormal bone subclinical and take care to avoid changes to bone deformities and find ways to treat them.

ELIGIBILITY:
Inclusion Criteria:

* Adult with type 1 or 2 diabetes with or without neuropathy

Exclusion Criteria:

* Pathology affecting bone metabolism:

  * abnormalities of phosphate metabolism proved biologically hepatic,
  * chronic alcoholism
  * renal insufficiency (creatinine clearance < 60 ml / min)
  * hyperthyroidism,
  * intoxication active smoking,
  * occlusive arteritis of lower limbs (IPS > IPS 1.2 or < 0.9)
* Treatment affecting bone metabolism (corticosteroids or glitazones for over 3 months in the year or bisphosphonates within 6 months)
* Known HIV positive serology
* Progressive, inflammatory disease (rheumatoid arthritis, ankylosing spondylitis, bowel inflammatory)

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-03-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07-10 (Actual)

PRIMARY OUTCOMES:
evaluate the MicroScanner, alterations quantitative and qualitative bone in the foot in patients with type 1 diabetes 2 with or without neuropathy | 18 month

SECONDARY OUTCOMES:
correlation involving bone and extension of neuropathy Assessment criteria associated with biological abnormalities qualitative and quantitative bone in diabetic subjects | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Boitard, MD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hotel Dieu, Paris, France